CLINICAL TRIAL: NCT04442724
Title: Bladder Fiducial Markers and Multiparametric-MRI (Mp-MRI) to Optimize Bladder Chemo-radiotherapy
Acronym: FMBRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Maurice M. Garcia, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2017-12-Garcia-FMBRT; 1R01CA201709-01 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer; Urinary Bladder Neoplasm; Urologic Neoplasms; Neoplasms; Urinary Bladder Diseases
Keywords: Fiducial marker; Fiducial marker guided technique
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms; Neoplasms; Urinary Bladder Diseases | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm - Bladder Chemo-Radiotherapy (Experimental): Fiducial marker placement & cystogram during resection surgery, followed by radiation planning CT scan, mpMRI, chemo-radiation treatment; mpMRI and/or surveillance cystoscopy at 3, 6, and 9 months post-treatment.
  Interventions: Procedure: Fiducial marker placement; Diagnostic Test: Multiparametric MRI (mpMRI)

INTERVENTIONS:
Procedure: Fiducial marker placement — placement of 24k gold fiducial markers surrounding the tumor site, at time of primary or re-staging bladder tumor resection
Diagnostic Test: Multiparametric MRI (mpMRI) — In this study, mp-MRI is defined as MRI that includes T1 & T2 weighted sequences, diffusion weighted sequences, and Dynamic contrast enhanced (DCE) MRI sequences.

SUMMARY:
The purpose of this study is to examine the usefulness of implanting small 24-K gold fiducial markers around a bladder tumor site, so that a Radiation Oncologist can identify the original tumor location at the time of radiation treatment. Other goals of the study include assessing whether a new MRI imaging technology can help with detection of bladder cancer earlier and more accurately when evidence of bladder cancer is not visible by scope.

DETAILED DESCRIPTION:
This study of fiducial markers in patients with localized muscle-invasive bladder cancer will enroll patients electing bladder preservation with tri-modal therapy.

24-K gold fiducial markers will be endoscopically implanted around the tumor resection area to mark the location of the tumor site, into the bladder wall submucosa space under direct visualization via a coaxial needle. The markers are visible on all imaging modalities, including all available on-table imaging (e.g., portal and cone-beam CT) used for radiotherapy. Reliable fiducial marker placement within the bladder may have the potential to advance bladder-sparing management of localized muscle-invasive bladder cancer.

This study will examine the effectiveness of bladder-preserving multi-modal treatment of muscle-invasive bladder cancer with and without fiducial marker placement to guide radiotherapy targeting and to minimize collateral radiation. In addition, this study intends to verify the accuracy and report on the sensitivity and specificity of mp-MRI imaging to detect the presence and location of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of primary urothelial carcinoma of the bladder. Subjects with mixed histology are required to have a dominant traditional cell carcinoma (TCC) pattern.
* Clinical stage T2-T4a, Nx, M0 considered appropriate for, and electing to receive, chemoradiation of the bladder
* Planned TURBT as part of the normal course treatment, to take place prior to the initiation of chemo irradiation
* Adequate renal function: Serum creatinine < 2 mg/dL OR calculated creatinine clearance (CrCl) > 30ml/min
* Ability to understand and willingness to sign a written informed consent
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, during study participation, and for 90 days after study treatment discontinuation

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Subjects with primary TCC of the ureter, urethra, or renal pelvis, without TCC of the bladder, are not allowed
* Known distant metastatic disease (e.g. pulmonary or hepatic metastases)

  * Subjects with malignant lymphadenopathy in the abdomen or pelvis considered appropriate for radical cystectomy and lymphadenectomy with the goal of complete resection of all malignant disease are allowed
* Patients with bladder abnormalities that preclude safe placement of fiducial markers (i.e. abundant large diverticuli or cellules, active or recurrent urinary infection)
* Planned (or prior history of) definitive bladder irradiation
* Intravesical chemo- or biologic therapy within 6 weeks of first treatment
* Any planned neoadjuvant systemic immunotherapy. Note that prior bacille Calmette-Guerin vaccine (BCG) is not an exclusion
* Clinically significant active infection or uncontrolled medical condition that would preclude participation in study
* Pregnant or nursing women are excluded
* Previous malignancy other than TCC that, in the opinion of the treating investigator, is likely to interfere with protocol treatment
* Individuals with severe renal failure and cannot receive MRI contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Bladder volume differential | Baseline, after marker placement (anticipated to occur between study days 0-1)
  Change in bladder volumes targeted for high dose radiation (HDR) between the first (Baseline) dose volume histogram (DVH) without the fiducial markers present, compared to the second DVH made after placement of the fiducial markers

SECONDARY OUTCOMES:
Net dose radiation to collateral organs differential | Baseline, after marker placement (anticipated to occur between study days 0-1)
  comparison of a DVH (Dose Volume Histogram) made without the fiducial markers present, to the second DVH made with the fiducial markers present. This will be measured by net dose (Gy to area and/or volume) to collateral organs
Positive Predictive Value of Multiparametric-MRI (mp-MRI) | at the time of initial TURBT (Day 1), at the initial post-treatment surveillance cystoscopy (3 months post-treatment)
  percentage of actual positive sites among those predicted positive by mpMRI
Difference in alignment when markers are incorporated into the planning | Radiotherapy treatment period (Days 14-28)
  Difference in "on-table" patient alignment under the radiotherapy gantry (in millimeters, in X, Y and Z dimensions) when the patient is aligned daily based on conventional methods only (i.e. fiducial markers are not used for alignment), and when the patient is aligned based on the fiducial markers as the reference.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Garcia, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center (CSMC), Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Harvard School of Medicine/Massachusetts General Hospital (MGH), Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No